CLINICAL TRIAL: NCT06117137
Title: The Impact Of Sodium-Glucose Cotransporter 2 Inhibitors on Metabolic Dysfunction -Associated Steatotic Liver Disease In Patients With Type 2 Diabetes Mellitus
Brief Title: The Impact Of SGLT2 -I on Metabolic Dysfunction -Associated Steatotic Liver Disease In Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, George Esmat Roshdy, Assistant lecturer at internal medicine department faculty of medicine sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-10-06MD
Record Dates: First submitted 2023-10-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Fatty Liver, Nonalcoholic
Keywords: Sglt2-I; Metabolic associated steatotic liver disease; Type 2 diabetes mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Control group (stander treatment of Type 2 diabetes mellitus without SGLT2-I ) SGLT2-I groups (stander treatment of Type 2 diabetes mellitus plus SGLT2-I )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Experimental): Control group (stander treatment of Type two diabetes mellitus without SGLT2-I )
  Interventions: Drug: SGLT2 inhibitor
- Group dapa (Experimental): Dapa group: (stander treatment of type two diabetes mellitus plus Dapagliflozin)
  Interventions: Drug: SGLT2 inhibitor
- Group empa (Experimental): Group empagliflozin: stander treatment of type two diabetes mellitus plus empagliflozin
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Group empagliflozin: stander treatment of type two diabetes mellitus plus empagliflozin
  Group dapa:standard treatment of type 2 Diabetes mellitus and dapagliflozin
  Other Names: Empagliflozin ,Dapagliflozin

SUMMARY:
Study question 1:Could SGLT2-I improve hepatic fibrosis, steatosis, and inflammatory markers in type 2 diabetic patients with Metabolic associated steatotic liver disease Question 2:Which drug of SGLT2-I group is more effective in improving metabolic associated steatotic liver disease in type 2 diabetic patients?

DETAILED DESCRIPTION:
patients will be derived from Endocrine or Hepatology outpatient clinic and who were primarily visiting for management of type 2 diabetes and other comorbidities.

The effect of the SGLT2-I on metabolic associated steatotic liver disease patients with Type two diabetes mellitus will be a prospective, open-label, parallel-groups, randomized clinical study to examine the effect of different types of SGLT2-I (dapagliflozin, empagliflozin,) when included in the standard treatment of Type two diabetes mellitus versus standard treatment without SGLT2-I for 24 weeks based on a predefined computer-generated number with a 1:1 allocation that will be concealed in patients with Type 2 diabetes mellitus and Metabolic associated steatotic liver disease Patients will be treated with combination therapy metformin and/or sulfonylurea and/or dipeptidyl peptidase 4 (DPP-4) inhibitors and/or insulin (control group), for whom treatment with SGLT2-I plus standard treatment for type 2 diabetes. (SGLT2-I group) will be indicated due to poor diabetes control

- The patients will subsequently be classified and treated by the lines of diabetes therapy (based on randomization into SGLT2-I or control group).

Baseline assessment (First visit)

All patients before randomization will be subjected to :

Detailed medical history including:

Demographic characteristics, Medications for glycemic control Compliance on medications Duration of Diabetes and presence of any comorbidity Diabetes complications.

Detailed clinical examinations including:

Height, weight, waist circumference Systolic blood pressure and diastolic blood pressure. Body mass index (BMI) is calculated with division of weight (in kg) by square of height (in meters).

3 - Laboratory investigations: Plasma glucose level Glycated hemoglobin (HbA1c) Blood urea and serum creatinine, Serum uric acid, Total bilirubin (mg/dL) Alanine aminotransferase (units/L), Aspartate aminotransferase(units/L) Albumin (units/L) Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglyceride, Plasma non-HDL-cholesterol was simply calculated by following formula: total cholesterol- HDL cholesterol.

Uric acid to cholesterol ratio is calculated with division of serum uric acid by HDL cholesterol.

The Uric acid to non-HDL cholesterol ratio is measured by the following formula: uric acid/non-HDL cholesterol.

Hepatitis B surface antigen, anti-hepatitis C and HIV I and II antibodies. Urine analysis and Albumin-to-creatinine ratio Complete blood counts Monocyte to high-density lipoprotein cholesterol ratio Neutrophil to lymphocyte ratio Platelet to lymphocyte ratio Lymphocyte to monocyte ratio Neutrophil-percentage-to-albumin ratio ECG 4-Other investigations will be including: Abdominal ultrasonography (Liver & spleen size, portal vein diameter) 5- Non-Invasive Testing of Hepatic steatosis/fibrosis: Using vibration-controlled transient elastography (FibroScan), Study visits All participants will be instructed about potential adverse drug reactions. Each participant will be asked to document all the symptoms that they will experience during the study period, whether related to drug or not.

Compliance and adverse events will be assessed by a verbal questionnaire. In both groups, adjustment of diabetes treatment will be carried out based on self-monitored blood glucose at weeks 4 and 8 by telephone consultation.

All participants will be instructed to restrict simple carbohydrates (avoid simple sugars, reduce rice preparations) and fat intake (reduce butter, ghee).

All participants will be advised to exercise (brisk walk) for at least 45 min a day for at least 5 days a week.

Participants will return to the outpatient hepatology clinic for follow-up visits at weeks 12 and 24.

All the participants, at baseline and at week 12, will receive uniform lifestyle modification instructions in accordance with the standards of diabetes management Anthropometry, physical examination results and biochemical measurements will be recorded for each participant in week 24.

Biochemical measurements at follow-up

Venous blood samples will be taken at week 24 in the morning after participants had fasted overnight for 12 h and the samples will be analyzed on the same day at the center laboratory of the hospital for the previous variables.

Vibration controlled transient elastography (VCTE) parameters

Liver stiffness measurement (LSM) by VCTE (related to liver fibrosis) and controlled attenuation parameter (CAP; related to liver fat) will be measured using Fibroscan a trained hepatologist who will be blinded to the drug allocation, clinical data, and biomarker data.

Study group:

At the end of the study, all the patients will be classified according to Type of treatment Control group (stander treatment of Type 2 diabetes mellitus without SGLT2-I ) SGLT2-I groups (stander treatment of Type 2 diabetes mellitus plus SGLT2-I )

SGLT2-I group will be sub-grouped to Group dapagliflozin: stander treatment of Type 2 diabetes mellitus plus dapagliflozin Group empagliflozin: stander treatment of Type 2 diabetes mellitus plus empagliflozin

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥20 years old who will be:

  1. Diagnosed with type 2 diabetes since ≥6 months in accordance with World Health Organization criteria (22); and
  2. Present with glycated hemoglobin equal to or greater than 7% and less than 10% after at least three months of treatment with metformin monotherapy at the maximal tolerated dosage or sulfonylurea alone or in combination; and
  3. Diagnosed with Metabolic associated steatotic liver disease

     Exclusion Criteria:
* Diagnosis or signs of type 1 diabetes or non-diabetic patients
* Highly uncontrolled diabetes (HbA1c >86 mmol/mol [>10.0%])
* BMI ≥40 kg/m2
* Other causes of chronic hepatic steatosis (e.g., Hepatitis B virus ,Hepatitis c virus, autoimmune disease, Wilson disease, drugs, alpha one antitrypsin deficiency).
* Patients use of drugs known to cause hepatic steatosis (e.g., amiodarone, valproate, tamoxifen, methotrexate, steroids)
* Treatment with glucose-lowering drugs that influence liver fat, including thiazolidinediones, α-glucosidase inhibitors, sodium-glucose cotransporter 2 (SGLT2) inhibitors or any glucagon-like peptide-1 receptor agonists during the previous 3 months.
* Detection of biliary duct obstruction based on imaging studies.
* Patients with diagnosis of or clinical features that are suspected for another systemic disease that commonly causes liver disease.
* Patient with history of liver transplantation
* Evidence of cirrhosis (on basis of ultrasonography and MRI) or hepatocellular carcinoma (evidence on triphasic CT or MRI).
* Positive HIV test
* Treatment with vitamin E during the previous 3 months.
* Intolerance or allergy SGLT2-I or any other substance in the tablets.
* Contraindications to SGLT2-I use (history of acute or chronic pancreatitis or pancreatic cancer, or history of recurrent urinary tract or genital infections, current or previous gangrene).
* History of or presence of (as found at Visit 1) any clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
* Creatinine clearance <90 ml/min at screening (Cockcroft-Gault formula).
* Severe hepatic injury and/or significant abnormal liver function defined as aspartate aminotransferase >5× upper limit of normal (ULN) and/or alanine aminotransferase >5× ULN.
* Total bilirubin >2.0 mg/dl (34.2 μmol/l)\
* History of bariatric surgery or ongoing weight-loss diet (hypocaloric diet) or use of weight-loss agents unless the diet or treatment has been stopped at least 3 months before screening and that the patient has had a stable body weight (+/- 3 kg) during the 3 months before screening.
* Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results as judged by the investigator. This includes signs of liver disease other than non-alcoholic fatty liver disease that motivated further investigations or treatment based on clinical judgment.
* Drug abuse or alcohol abuse.
* Women who are pregnant, lactating or planning to become pregnant during the study period, or women of childbearing potential who are not using acceptable contraceptive methods. A woman is considered of childbearing potential if she is not surgically sterile or is less than 1 year since last menstrual period. Acceptable contraceptive methods will be combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion and vasectomized.
* Any other condition the investigator believed would interfere with the patient's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the patient at undue risk.
* Any blood donation/blood loss >500 ml during the 3 months prior to Visit 1 or during the study.
* Patients with active malignancy
* Patients with established hemolytic disease
* Refused to consent to this study.
* The patient will be excluded from the study after the randomization if the second compound of combination therapy is inconsistent with the standard of medical care in diabetes -2022.
* Patient use of anti-inflammatory medications or corticosteroids during the observational period
* Missing the follow up.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
Number of participants with tight controlled diabetes melitus | 6 months
  Measurement of glycated hemoglobin, random blood sugar,fasting blood sugar

SECONDARY OUTCOMES:
Number of participants with changing in liver stiffness measurement (LSM in kPa) measured by vibration-controlled transient elastography | 6 months
  Fibroscan before and after 6 months duration of treatment
Number of participants with changing Liver and spleen size | 6 months
  Abdominal ultrasound
Number of participant with changing in inflammatory biomarkers | 6 months
  Measurement of Monocyte to high-density lipoprotein cholesterol ratio Neutrophil to lymphocyte ratio Platelet to lymphocyte ratio Lymphocyte to monocyte ratio Neutrophil-percentage-to-albumin ratio

IPD SHARING:
Plan to Share IPD: No